CLINICAL TRIAL: NCT06535828
Title: AIM4 AI and Mechanistic Modeling in Molecular Medicine
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn No Participants Enrolled
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Phase One Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0886; NCI-2024-06520 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Molecular Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AI and mechanic modeling: Participants with advanced/unresectable stage III or metastatic HR+ breast cancer with progression on a CDK4/6i and an AI will be eligible for study participation. The key action in this study will be the acquisition and analysis of tumor and blood for selection of standard of care systemic therapy. Tumor and blood will also be obtained at the time of disease progression to provide critical data for reverse translational model building. This will also provide insight into mechanisms of resistance for the administered standard of care therapy that can be used for future models to optimize selection of next-line therapy.
  Interventions: Device: AI and mechanic modeling

INTERVENTIONS:
Device: AI and mechanic modeling — The data collected from research tests on your blood and tumor samples will be used to develop an AI model for treatment selection.

SUMMARY:
To assess for potential pitfalls and to assess the feasibility of the approach of analysis of new tumor biopsies for selection of standard of care treatment selection in patients with metastatic hormone receptor positive breast cancer who have developed disease progression on 1st line endocrine therapy combined with a CDK4/6 inhibitor.

DETAILED DESCRIPTION:
Primary Objective To assess the feasibility and utility of tumor evaluation to aid in selection of standard of care therapy for patients with hormone receptor positive (HR+) /HER2- advanced/metastatic breast cancer.

Secondary Objectives

* Accrual Rate (AR)
* Clinical Benefit Rate (CBR)
* To compare progression free survival (PFS) based on concordance with recommended treatment
* Duration of Response (DoR)
* Therapy Acceptance Rate (TAR)

ELIGIBILITY:
Inclusion Criteria:

* Eligibility will be evaluated by the study team according to the following criteria. Subjects must meet all of the inclusion and none of the exclusion criteria to be registered to the study. Study treatment may not begin until a subject is registered.
* Patients must have histologically confirmed, advanced/unresectable stage III or metastatic hormone receptor positive, HER2 breast cancer. Hormone receptor positive is defined as estrogen receptor >= 10% and/or progesterone receptor >=10%. Her2 negative per American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP) guidelines.
* Patient must have disease progression during or after CDK4/6 inhibitor (CDK4/6i) combination treatment with an aromatase inhibitor (AI) meeting one of the following criteria.
* Disease progression on treatment with a CDK4/6i and AI as 1st line endocrine therapy for advanced/metastatic breast cancer.
* Disease progression on or following treatment with a CDK4/6i in the adjuvant setting for early-stage breast cancer.
* Age ≥ 18 years.
* ECOG performance status of ≤2.
* Patient must have at least one lesion amenable to percutaneous core biopsy that is not a purely sclerotic bone lesion.
* Patient must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.

Exclusion Criteria:

* Pregnant or lactating women.
* Prior treatment with capecitabine, phosphoinositide 3 kinase (PI3K) inhibitor, mechanistic target of rapamycin (mTOR) inhibitor, protein kinase B (Akt) inhibitor, selective estrogen receptor degrader (SERD), or HER2-targeted therapy, including neratinib.
* Known and untreated, or active, brain or leptomeningeal metastases. Subjects with previously treated central nervous system (CNS) metastases may be enrolled in the study if they do not require systemic steroids, do not have seizures ort uncontrolled neurological symptoms, and have stable disease confirmed by radiographic assessment within at least 4 weeks prior to enrollment.
* History of malignancies other than adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥3 years.
* Platelet count < 100,000/microliter or INR >1.5.
* Life expectancy <1 year.
* Participants who are consented to participate in the clinical trial, who do not meet one or more criteria required for participation in the trial during the screening procedures, are considered screen failures. Records of participant screening to include screen failures will be maintained by the clinical research team. There is no role for re-evaluation and re-screening of patients once they have deemed to be a screen failure.
* Both men and women of all races and ethnic groups are eligible for this trial, although women comprise the majority of breast cancer patients and will be largely represented in this trial. Males are estimated to make up 1% of total breast cancer cases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Azadeh Nasrazadani, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org